CLINICAL TRIAL: NCT04150939
Title: Cryoablation Challenge Evaluated in Adaptive-Immune Resistance (CEDAR)
Brief Title: Cryoablation for the Treatment of Metastatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0502; NCI-2019-07100 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0502 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy, Needle; Biopsy, Large-Core Needle; Cryosurgery; Adjuvants, Immunologic; Immunologic Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (cryoablation) (Experimental): Beginning 1 week prior to the next scheduled standard of care immunotherapy infusion, patients undergo core biopsy of the lesion to be ablated and a non-ablated lesion and also undergo cryoablation. Patients undergo a mandatory second core biopsy of the non-ablated lesion at 4 weeks after cryoablation.
  Interventions: Procedure: Core Biopsy; Procedure: Cryosurgery; Drug: Immunotherapeutic Agent

INTERVENTIONS:
Procedure: Core Biopsy — Undergo core biospy
  Other Names: core needle biopsy
Procedure: Cryosurgery — Undergo cryoablation
  Other Names: Cryoablation; cryosurgical ablation
Drug: Immunotherapeutic Agent — Receive standard of care immunotherapy
  Other Names: Biological Response Modifier; Biomodulators; BRM; Immune Mediators; Immune Modulators; Immune Regulators; Immunomodulating Agent; Immunomodulators; Immunomodulatory Agent; Immunopotentiators; Immunotherapy Agent

SUMMARY:
This interventional trial studies the effectiveness of adding cryoablation treatment in patients who are receiving standard of care immunotherapy to treat cancer that is has spread to other parts of the body (metastatic). Cryoablation uses a probe that freezes the tissue around the tumor to try to kill the cancer cells. Using cryoablation to treat cancerous lesions may help to kill the cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of cryoablation on adaptive resistance to immunotherapy in metastatic cancer patients.

SECONDARY OBJECTIVES:

I. To assess additional efficacy response to treatment. II. To assess the safety and tolerability of cryoablation in this population. III. To compare the radiologic response of ablated and non-ablated lesions using Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST) and RECIST 1.1.

IV. To assess the immune effect of cryoablation on the non-ablated lesion using pre- and post-treatment biopsies.

EXPLORATORY OBJECTIVE:

I. To evaluate the immune microenvironment and systemic changes as a result of cryoablation with the goal of biomarker discovery.

OUTLINE:

Beginning 1 week prior to the next scheduled standard of care immunotherapy infusion, patients undergo core biopsy of the lesion to be ablated and a non-ablated lesion and also undergo cryoablation. Patients undergo a mandatory second core biopsy of the non-ablated lesion at 4 weeks after cryoablation.

After completion of study, patients are followed up for 12 months after cryoablation and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically confirmed metastatic cancer and be receiving standard of care immunotherapy (PD1/PD-L1 based therapy alone or in combination with other agents (i.e. chemotherapy, targeted therapy, CTLA-4 agent)
* Patient must have had >= 70% of planned dosing schedule of PD1/PD-L1 based therapy over the prior treatment period, defined as the previous 3 months

  * For example, the expected number of doses in three months for nivolumab dosed every 2 weeks would be 6 infusions. If the patient were able to receive 5 out of the 6 doses (83% of planned dosing schedule), they would be eligible for the protocol. If the patient received only 4 out of the planned 6 doses (67% of planned dosing schedule), they would be ineligible for the protocol
* Immunotherapy treatment must have been given within the last 4 weeks without the need for systemic steroid therapy (excluding physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent)
* Patient must have demonstrated prior clinical benefit to PD1/PD-L1 based therapy followed by progression as defined by RECIST1.1: 1) partial response (PR) or complete response (CR) by RECIST1.1 (then progression by RECIST1.1) 2) stable disease (SD) x 6 months (then progression by RECIST1.1)
* Patient must have at least two lesions not previously treated with loco-regional therapy (including external beam radiation, embolization (bland or chemo), Y90, prior ablation (i.e. microwave, radiofrequency ablation, cryoablation, irreversible electroporation) that can be accurately measured in at least one dimension (longest diameter to be recorded) as >=10 mm with spiral computed tomography [CT] scan or >= 20 mm with magnetic resonance imaging [MRI])
* Patient must not have a contraindication to continuing on their current immunotherapy dose regimen for at least 3 months post-cryoablation
* All lines of prior therapy accepted. Patients with resections of metastatic disease will be included
* Life expectancy of greater than 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Total bilirubin < 1.5 X institutional normal limits (subjects with known Gilbert syndrome are eligible with total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal
* Creatinine within normal institutional limits OR - creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, tubal ligation or hysterectomy)
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. Women >= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, tubal ligation or hysterectomy)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior immune-related drug toxicity related adverse events that have not recovered to baseline or grade 1 (alopecia excluded)
* Patient may not be receiving any other investigational agents
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]) that require treatment with a disease modifying agent.

  * The following are exceptions:

    * Patients with the above disorders may be considered upon principal investigator (PI) review and allowance (i.e. patient had an autoimmune or inflammatory disorder but despite the diagnosis has been tolerating immunotherapy)
    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
* Current use of immunosuppressive medication including for the treatment of severe immune toxicity related to PD1/PD-L1 based therapy that precludes further treatment with immunotherapy agents. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of active primary immunodeficiency
* Pregnant or nursing women; women of childbearing potential unless using effective contraception as determined by the investigator
* Receipt of a live vaccine within 30 days of study entry
* Any concurrent hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (e.g. hormone replacement therapy) is acceptable
* Patient who does not have lesions suitable for biopsy and cryoablation or measurable disease (non-ablated lesion)
* The lesion being considered for cryoablation must not have undergone prior local therapy (radiation treatment, embolization (including bland embolization or chemoembolization), yttrium therapy, prior ablation of any modality (microwave, radiofrequency ablation, cryoablation, irreversible electroporation)
* Patient with symptomatic central nervous system (CNS) brain metastases, craniospinal metastases, uncontrolled seizure disorder, or active neurological disease. Patients presenting with brain metastases must be asymptomatic or treated and stable off steroids and anti-convulsants for at least 1 month prior to study treatment
* Patient with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Contraindication to enhanced magnetic resonance imaging (MRI) or computerized tomography (CT) imaging (according to patient characteristics and investigator decision)
* Absolute contraindication or known untreatable allergic reactions to contrast media agents
* History of allogenic organ transplantation
* Known active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive hepatitis B [HBV] surface antigen [HBsAg] result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Best objective response (complete response or partial response) | Up to 12 months post cryoablation
  Will be determined by Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST). Best objective response will be measured by the proportion of patients who achieve complete response (CR) + partial response (PR). The proportion of patients in the efficacy evaluable population who respond (i.e., have a best response of CR or PR) will be estimated along with the corresponding 95% confidence interval, using the Clopper-Pearson exact method.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 2 years
  Will be determined by iRECIST. PFS will be calculated and plotted by Kaplan-Meier methods.
Time to progression (TTP) | Up to 2 years
  Will be determined by iRECIST. TTP will be calculated and plotted by Kaplan-Meier methods
Time to progression on a ablated versus non-ablated basis | Up to 2 years
  Ablated lesions time to progression will be determined b iRECIST and RECIST 1.1. Non-ablated lesion time to progression will be determined by iRECIST and RECIST 1.1. TTP will be calculated and plotted by Kaplan-Meier methods.
Disease control rate (CR + PR + stable disease [SD]) | Up to 2 years
  Descriptive statistics will summarize disease control rate by iRECIST.
Duration of stable disease | Up to 2 years
  Descriptive statistics will summarize duration of stable disease by iRECIST.
Duration of response | Up to 2 years
  Descriptive statistics will summarize duration of response by iRECIST.
Incidence of adverse events (AEs) | Up to 2 years
  AEs will be graded and categorized according to Common Terminology Criteria for Adverse Events (CTCAE) version 5. Counts and percentages of patients experiencing each adverse event as well as any grade 3 or higher event will be summarized.
Overall survival (OS) | From the date of study entry until death from any cause, assessed up to 2 years
  OS will be calculated and plotted by Kaplan-Meier methods.
Changes in T-effector cell populations | Baseline up to 12 months post cryoablation
  Will use a paired t test to determine if there is a difference in pre- and post immune cryoablation therapy in T-effector cell populations; T-regulatory populations; CD4 subsets; B cell populations; dendritic and macrophage populations. Will use scatterplots to demonstrate correlation between immunologic markers obtained in peripheral blood versus those obtained at the tissue level. A Pearson correlation will be estimated to describe the level of association.

OTHER OUTCOMES:
Immune parameters | Up to 2 years
  Will assess various immune parameters in blood and tissue, including changes in immune cell composition and peripheral blood samples. Will use scatterplots to demonstrate correlation between immunologic markers obtained in peripheral blood versus those obtained at the tissue level. A Pearson correlation will be estimated to describe the level of association.

CONTACTS AND LOCATIONS:
Overall Officials: Alda L Tam, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT04150939/ICF_000.pdf